CLINICAL TRIAL: NCT02391207
Title: Hepatic Vein-sparing Hepatectomy for Colorectal Liver Metastases at the Caval Confluence: Validation on Intention-to-treat Analysis of a IOUS-guided Approach
Brief Title: Hepatic Vein-sparing Hepatectomy for Colorectal Liver Metastases at the Caval Confluence
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, Guido Torzilli, MD, PhD, FACS, Professor of Surgery, Director Department of Hepatobiliary & General Surgery, University of Milan, Humanitas Research Hospital, Rozzano, Milan, University of Milan
Other Study IDs: HV-SparingHx
Record Dates: First submitted 2015-03-07; First posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Secondary Malignant Neoplasm of Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients having at least one CLM: Hepatic vein-sparing hepatectomy guided by intraoperative ultrasonography
  Interventions: Procedure: Hepatic vein-sparing hepatectomy

INTERVENTIONS:
Procedure: Hepatic vein-sparing hepatectomy — HV detachment, partial resection and section on the basis of HV-CLM relationship

SUMMARY:
Major hepatectomies are generally selected for tumors involving the hepatic vein (HV) at the caval confluence (CC). As alternative, HV reconstruction has been proposed. The present study aimed to evaluate the feasibility and safety of a HV-sparing policy guided by intraoperative ultrasonography (IOUS) in a cohort of patients having at least one colorectal liver metastasis (CLM) in contact with a HV at CC. HV section can be avoided in the large majority of cases thanking to CLMs detachment or to HV partial resection or reconstruction: this policy seems feasible, safe, reduces the need of major hepatectomies, and oncologically provides an adequate local control.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of at least one CLM in contact with HV at caval confluence and HV patency at preoperative imaging
* at least 6 months of follow-up after surgery

Exclusion Criteria:

* suspected or ascertained thrombosis or full tumoral involvement of HV at preoperative imaging
* portal pedicle infiltration and/or thrombosis
* unresectability at laparotomy for any extra-hepatic or intrahepatic reason not related to tumor-vessel relations

Ages: 28 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patiens undergoing hepatectomy for primary and secondary liver tumors
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
the safety of HV-sparing surgery in terms of operative mortality and morbidity | within 30-90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Guido Torzilli, MD,PhD,FACS, Study Director — Department of Hepatobiliary and General Surgery, University of Milan, Humanitas Research Hospital, Rozzano, Milan, Italy; Fabio Procopio, MD, Principal Investigator — Department of Hepatobiliary and General Surgery, University of Milan, Humanitas Research Hospital, Rozzano, Milan, Italy
Locations (1):
- Department of Hepatobiliary and General Surgery, Humanitas Research Hospital, University of Milan, Rozzano, Milan, Italy